CLINICAL TRIAL: NCT06130371
Title: Stress, Inflammation and Neuroimaging in Major Depressive Disorder as Compared to Premenstrual Dysphoric Disorder
Status: Recruiting | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Dr. Ann-Christine Ehlis, Leader of the Research Group Psychophysiology & Optical Imaging Techniques, University Hospital Tuebingen
Other Study IDs: 340/2023BO2
Record Dates: First submitted 2023-09-05; First posted 2023-11-14 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: MDD; PMDD
Keywords: MDD; PMDD; Stress; Inflammation; Cytokines; fMRI; MIST
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- major depressive disorder group: female MDD patients with moderate levels of depressive symptoms, mostly recruited from psychotherapist offices and the outpatient clinic of the university.
- premenstrual dysphoric disorder group: female participants suffering from premenstrual dysphoric disorder, as confirmed by prospective ratings of premenstrual symptoms via an app during two consecutive menstrual cycles.
- healthy controls: healthy controls

SUMMARY:
Premenstrual dysphoric disorder (PMDD) is a sex-specific depressive disorder where depressive symptom severity drastically changes in relation to menstrual cycle phase. It is characterized by late luteal phase symptoms of affective lability, irritability, depressed mood, and anxiety. A lot remains unclear and further studies are needed in order to improve the understanding of PMDD and to differentiate it from major depressive disorder (MDD). To date, and in contrast to MDD, the neural correlates of PMDD have been sparsely and poorly investigated. The aim of this study is therefore to investigate the neural correlates of PMDD as compared to MDD and to relate them to stress reactivity. Therefore, three groups of naturally cycling women will be investigated and compared, namely (1) women with MDD, (2) women with PMDD, and (3) healthy control women.

Stress and HPA axis activity are assumed to play a crucial role in the development of many mental disorders, including MDD. How stress reactivity and HPA axis activity are connected to PMDD still needs to be investigated. Furthermore, the HPA axis can affect or suppress the activity of the hypothalamic-pituitary-gonadal (HPG) axis, which is involved mainly in the reproductive, but also the immune system, making it an important candidate for the investigation of sex-specific differences in stress reactivity.

There are sex-specific differences in stress reactivity, but also in the prevalence of stress-related diseases. Women are twice as likely to suffer from depression than men and the first onset of MDD usually peaks during the reproductive years. As to why these differences exist, a recent theory suggests that ovarian hormone fluctuations function as modulators of women's susceptibility to stress and that altered reactivity to stressors during different cycle phases plays a role in the etiology of depressive disorders. This hypothesis extends the Social Signal Transduction Theory of Depression which first and foremost relates depression to inflammation. They postulate a critical role of cytokines for understanding the pathogenesis of depression. Therefore, ovarian hormone fluctuations, but also inflammation in regard to MDD and PMDD and stress reactivity will be investigated in this study.

DETAILED DESCRIPTION:
In the proposed study the investigators aim to investigate in more detail how women with MDD and women with PMDD differ in their stress response from healthy women. The investigators are directly comparing three groups of 1) women with MDD, 2) women with PMDD and 3) healthy women. All women will be measured in two different cycle phases to disentangle the effects of the menstrual cycle on stress reactivity. Furthermore, including inflammatory markers will help to shed light on the connection between stress, depressive disorders and the immune system.

The overall aim of this study is to elucidate the influence of stress on inflammation as well as on brain function in women with MDD in contrast to PMDD. Therefore, the behavioral, neural, immunological, and endocrine profiles of women with MDD as well as women with PMDD will be compared to the ones of naturally cycling women. The goal is to delineate the psychobiological characteristics of reproductive states and mental disorders. The results will provide the basis to develop more targeted treatments in the framework of precision medicine.

Open questions:

1. How do women with MDD, women with PMDD, and healthy women differ in their stress reactivity on a neural level, as measured by fMRI activity?
2. How do women with MDD, women with PMDD, and healthy women differ in their stress reactivity in their HPA axis response, as measured via cortisol levels?
3. How do women with MDD, women with PMDD, and healthy women differ in their stress reactivity on an immunological level, as measured by inflammation markers?

The investigators hypothesize that after an acute psychosocial stressor,

1. women with MDD show hypoactivation in the CCN, especially so in the left DLPFC, when compared to healthy controls. For women with PMDD, this effect might be pronounced only when tested in the symptomatic, meaning the late luteal menstrual cycle phase.
2. women with MDD have higher cortisol levels than healthy controls but show a blunted stress response. As there are no studies on cortisol reactivity in women with PMDD, it is unclear how they will react to stress compared to healthy and MDD women.
3. women with MDD have higher inflammatory markers (such as IL-6 and TNF-alpha) when compared to healthy controls. For women with PMDD the investigators also expect higher inflammatory markers than in healthy controls.

This combined neuroimaging and stress study will investigate naturally cycling women with MDD (n = 25), PMDD (n = 25) and matched healthy control women (n = 25). All participants will be exposed to the Montreal Imaging Stress Task (MIST), a stress induction task during neuroimaging using fMRI. In order to disentangle the influence of the menstrual cycle, within a randomized design, one session will take place during the mid-follicular phase and one during the late-luteal phase of the menstrual cycle. Besides assessing heart rate variability as a measure of stress, the investigators will obtain cortisol from saliva and hair samples, as well as steroids (e.g., progesterone, estrogen, and ALLO) and inflammation markers from blood samples (e.g., adipokines, IL-1, IL-6, and TNF-alpha).

The investigators plan to assess 75 women to compare women with MDD to women with PMDD and healthy women. In total, the following samples will be recruited:

* Group 1: 25 women with MDD
* Group 2: 25 women with PMDD
* Group 3: 25 healthy women

If subjects qualify for the current study, the investigators will invite them to the laboratory (T0) where they will give written, informed consent. Subsequently, the investigators will perform a standardized clinical interview to screen for mental disorders (SCID-5-CV). Participants will also be informed about the study process and the data analysis. After the interview, they will receive a password-protected link provided by email to assess, among others, depressive symptoms, personality traits, gender identity and norms, sexual health, state and trait anxiety, and verbal intelligence using questionnaires. Participants will also be asked to report their average cycle length. Participants then will be divided into two groups, where Group A has their first MRI session in the mid-follicular phase (before ovulation) and the second MRI session in the late-luteal phase (after ovulation), and Group B has the first MRI session in the late-luteal phase and the second MRI session in the mid-follicular phase. MRI sessions will be scheduled according to self-reported beginning of menses and self-reported average cycle length.

For the PMDD group, PMDD diagnosis has to be confirmed by daily, prospective ratings of premenstrual symptom severity during two consecutive cycles as this is an official criterion for the disorder in the DSM-5. For this the smartphone app m-path will be used. They will be asked daily about their premenstrual symptoms with the Daily Record of Severity of Problems Questionnaire (DRSP) that takes about 3 minutes per day.

At the beginning and the end of the MRI sessions T1 and T2, a blood draw of 30 ml will be performed by medically trained personnel. After ensuring that all requirements to take part in an MRI study are met, the participants will be put into the MRI, and the MIST will be applied. Throughout the session, saliva samples will be taken six times for the measurement of salivary cortisol: once at arrival, once before the MIST, 40 minutes after the MIST, 60 minutes after the MIST and 120 minutes after the MIST. Additionally, at both MRI sessions, hair samples are collected to record the cumulative cortisol secretion of the past three months (= 3cm hair). At the end of the last measurement day (T2), participants will be informed about the exact goals of the study and will have to sign a final consent form that their data can be used after full disclosure of the goals.

Montreal Imaging Stress Task In the Montreal Imaging Stress Task (MIST), a frequently used performance-based stress paradigm, arithmetic tasks are presented to generate increased cognitive workload and thus performance demands. The arithmetic tasks must be solved either without time pressure and social evaluation (control condition) or with time pressure and social evaluation (stress condition). Before entering the fMRI scanner, arithmetic tasks are practiced on a computer in an approximately 3-minute training session, in which task difficulty is determined for the fMRI measurement. In total, the MIST lasts about 20 minutes.

MRI measurements will be performed at the 3T PRISMA scanner located at the Department of Psychiatry and Psychotherapy, University Hospital Tübingen. On each measurement day, all participants will undergo the MIST, a resting-state scan, an anatomical scan and a diffusion tensor imaging (DTI) scan. For the resting-state scan (approx. 8 min), a low-TR multi-band echo-planar-imaging (EPI) sequence will be applied. Participants will be instructed to keep their eyes open while they are watching the Inscape movie that was specifically designed to improve imaging at rest. The anatomical scan (approx. 8 min) will be acquired using an MPRAGE (3-D Magnetization Prepared Rapid Gradient Echo) sequence consisting of 160 sagittal slices. Lastly, the DTI scan (approx. 8 min) will be performed. All MR parameters will be established with experts from the radiology department.

Determination of stress markers in saliva and hair. Biological stress markers are regarded as so-called "objective" stress measures which, in addition to subjective stress parameters, represent further facets of the multidimensionality of stress. While saliva samples can represent physiological acute stress reactions or characteristic circadian rhythms, hair samples represent the retrospective recording of cumulative cortisol secretion over a period of several months. In the course of the laboratory measurement, the investigators will repeatedly collect saliva samples in order to trace the stress reaction (i.e., increase in cortisol). Due to the circadian rhythm, the laboratory measurement takes place between 15.00 and 20.00 in the afternoon only on workdays. Additionally, one hair sample per MRI measurement is collected by cutting a small strand of hair as close to the scalp as possible as a marker for chronic stress.

Blood samples for hormones and epigenetics. For measuring, among others, estradiol, progesterone, allopregnanolone and testosterone, as well as inflammation markers (such as adipokines, interleukines, and TNF-alpha), ethylenediaminetetraacetic acid (EDTA) blood samples will be taken after the MRI sessions. In addition to the phenotypic characterization, all participants will provide EDTA-blood samples for epigenetic analyses which will be sent to the Department of Psychiatry and Psychotherapy, Research Group Molecular Psychiatry (Head: Prof. Dr. Vanessa Nieratschker) for storage and analysis. Methylation changes will be studied in peripheral blood due to the accessibility of the study material in living humans. The investigation of brain material of living human participants for epigenetic processes is unrealistic. As a similar differential methylation in peripheral blood as in the brain has been demonstrated for the candidate genes under investigation in this study, the investigators consider blood as an adequate surrogate material, reflecting the situation in the brain. Furthermore, epigenetic factors influence the psychophysiological stress response and can thus explain interindividual differences found within the current study.

ELIGIBILITY:
Inclusion Criteria:

* Women,
* age between 18 and 40 years (no menopausal women),
* regular menstrual cycles (25-31 days),
* normal body mass index (18-35 kg/m2),
* German language fluency

Exclusion Criteria:

* any neurological or mental disease (only for healthy participants)
* hormonal, metabolic or chronical diseases
* pregnancy
* women who gave birth or were breastfeeding within the last year
* women with any kind of steroid hormonal treatment
* oral contraceptive treatment in the last three months
* psychotropic treatment, only if regular
* engagement in competitive sports
* shift work

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be recruited by newspaper/social media advertisements, e-mails ("Rundmail") and posting notices ("Aushänge") at different places at the University Hospital Tübingen as well as the University of Tübingen and in social networks.
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2024-01-04 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
neural stress reactivity / activation of the CCN (cognitive control network) during stress-related tasks | during the MIST (20 minutes)
  activity in stress-circuits of the brain, especially DLPFC activity
stress-related cortisol reactivity | five cortisol measurements at MRI arrival, before the MIST, 50 minutes after the MIST, 70 minutes after the MIST, 120 minutes after the MIST
  cortisol level change in saliva between before and after the MIST
TNF-alpha in response to stress-related task | blood sample before and after the MIST (approx. 120 minutes)
  TNF-alpha in blood before / after the MIST
CRP in response to stress-related task | blood sample before and after the MIST (approx. 120 minutes)
  CRP in blood before / after the MIST
IL-6 in response to stress-related task | blood sample before and after the MIST (approx. 120 minutes)
  IL-6 in blood before / after the MIST
activity of parasympathetic nervous system (PNS) in response to stress-related task | change of RMSSD in relation to HRV during MIST (20 minutes)
  RMSSD (Root Mean Square of Successive Differences) of HRV
activity of parasympathetic nervous system (PNS) in response to stress-related task | change of pNN50 of HRV during MIST (20 minutes)
  pNN50 of HRV
activity of sympathetic nervous system (SNS) | change of skin conductance during MIST (20 minutes)
  skin conductance: galvanic skin response
chronic stress | measured at the first MRI and 2 weeks later at the second MRI
  cortisol in hair

SECONDARY OUTCOMES:
different levels of inflammation in Major Depressive Disorder, Premenstrual Dysphoric Disorder and Healthy Controls | Baseline (T1)
  ANOVA for different levels of CRP in different groups (PMDD, MDD, control)
different levels of inflammation in Major Depressive Disorder, Premenstrual Dysphoric Disorder and Healthy Controls | Baseline (T1)
  ANOVA for different levels of IL-6 in different groups (PMDD, MDD, control)
different levels of inflammation in Major Depressive Disorder, Premenstrual Dysphoric Disorder and Healthy Controls | Baseline (T1)
  ANOVA for different levels of TNF-alpha in different groups (PMDD, MDD, control)
changes in stress-reactivity induced by varying levels of sex hormones | MIST at T1 (follicular) and T2 (luteal phase) (2 weeks)
  ANOVA for cortisol reactivity between different cycle phases (luteal phase, follicular phase)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Fallgatter, Prof. Dr., Principal Investigator — Universitätsklinikum Tübingen, Klinik für Psychiatrie und Psychotherapie
Locations (1):
- University Hospital Tübingen, Klinik für Psychiatrie und Psychotherapie, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No